CLINICAL TRIAL: NCT05151861
Title: Withdrawal of Pharmacological Treatment in Patients Responding to Cardiac Resynchronization Therapy: Open and Randomized Study
Brief Title: Withdrawal of Pharmacological Treatment in Patients Responding to Cardiac Resynchronization Therapy:
Acronym: REMOVE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IMIB-RMV-2021-02
Record Dates: First submitted 2021-11-12; First posted 2021-12-09 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Complete removal of pharmacological treatment
  Interventions: Other: Complete removal of pharmacological treatment
- Control (Active Comparator): Maintenance of pharmacological treatment
  Interventions: Drug: Control

INTERVENTIONS:
Other: Complete removal of pharmacological treatment — Removal of treatment
  Arms: Experimental
Drug: Control — Maintenance of pharmacological treatment
  Arms: Control

SUMMARY:
The purpose of this randomized trial is to investigate the effect of the complete removal of pharmacological treatment in patients responding to cardiac resynchronization therapy with recuperated LVEF in terms of imaging parameters (changes in LVEF and LV volume), as well as, clinical parameters that translate into worsening of heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with a CRT device for at least one year due to the presence of LBBB and LVEF <40% of non-ischemic origin
2. Current LVEF ≥50% and normal volumes in two consecutive echocardiographic studies, separated at least 3 months, and the last one performed in the previous 6 months.
3. Normally functioning CRT device with stimulation> 95%.
4. NYHA functional class I-II.
5. Absence of admissions for HF in the last year.
6. NT-proBNP <450pg/ml in sinus rhythm and <900pg/ml in patients with atrial fibrillation, in the previous 6 months.
7. Pharmacological treatment with beta-blockers, ACEIs/AIIRA/RNAI with or without MRA.
8. Older than 18 years.
9. Patients who have given their informed consent in writing.

Exclusion Criteria:

1. Previous episode of sustained ventricular tachycardia/recovered sudden death/appropriate shock (in the case of a patient with an implantable cardioverter-defibrillator associated with CRT).
2. Uncontrolled arterial hypertension (figures> 140/90 mmHg).
3. Need to use beta-blockers at the medical discretion for other indications such as heart rate (HR) control in atrial fibrillation (in the absence of ablation of the atrioventricular node) or to control other supra or ventricular arrhythmias.
4. Severe valve disease.
5. Diabetic or hypertensive with microalbuminuria or proteinuria.
6. Renal failure with creatinine clearance <30ml/min/1.73m2.
7. Fertile women who are neither using contraceptives nor surgically sterilized; pregnant or lactating women.
8. Patients are currently participating in a clinical trial or have participated in the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-12-03 (Actual); Primary Completion 2022-11-15 (Estimated); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
1. A reduction in LVEF (Left ventricular ejection fraction) of more than 10% | Up to 48 weeks
  Number of patients with echocardiographic studies
2. An increase >15% in the VTSVIi (The end-systolic volume of the indexed left ventricle) to the previous one and in a range higher than the normal value | Up to 48 weeks
  Number of patients with echocardiographic studies
3. Clinical evidence of HF (Heart Failure) based on a global assessment, both clinical and analytical, together with the need to increase the dose of diuretics, as adjudicated by the research team. | Up to 48 weeks
  Number of patients with echocardiographic studies

SECONDARY OUTCOMES:
total mortality, (Number ) | Up to 48 weeks
  Total Number
Cardiovascular mortality, | Up to 48 weeks
  Total Number
Unplanned hospital admission or emergency room visit for HF (Heart Failure) | Up to 48 weeks
  Total Number
Unplanned hospital admission or emergency room visit for sustained atrial or ventricular arrhythmias (>30 seconds). | Up to 48 weeks
  Total Number
Changes with respect to baseline levels of BP (Blood pressure ) | Up to 48 weeks
Changes with respect to baseline levels of HR figures. (heart rate) | Up to 48 weeks
Change from baseline LVEF | Up to 48 weeks
Change from baseline left ventricular end-diastolic volume (VTDVIi) | Up to 48 weeks
Change from baseline body surface indexed left atrium volume (VAIi) | Up to 48 weeks
Changes from baseline in global longitudinal strain (GLS).GLS is a simple parameter that expresses longitudinal shortening as a percentage (change in length as a proportion to baseline length). | Up to 48 weeks
Changes in the quality of life questionnaires according to The Minnesota Living with Heart Failure (MLHFQ) scales. | Up to 48 weeks
  The response options range from 0, which indicates unaffected HRQL, to 5, which indicates the maximum impact on HRQL.
Changes in the quality of life questionnaires according to The Kansas City Cardiomyopathy Questionnaire (KCCQ) scales. | Up to 48 weeks
  The KCCQ is a 23-item (15 question) self-administered questionnaire designed to quantify physical limitations, symptoms (frequency, severity and recent change over time), social limitations, self-efficacy, and quality of life.As described, all KCCQ scores are scaled from 0 to 100 and frequently summarized in 25-point ranges, where scores represent health status as follows: 0 to 24: very poor to poor; 25 to 49: poor to fair; 50 to 74: fair to good; and 75 to 100: good to excellent.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco José Pastor Pérez, MD, Principal Investigator — HCUVA
Locations (1):
- Hospital Clínico Universitario Virgen de la Arrixaca, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pastor-Perez FJ, Garrido-Bravo IP, Penafiel-Verdu P, Fernandez-Villa N, Manzano-Fernandez S, Oliva-Sandoval MJ, Perez-Martinez MT, Caro-Martinez C, Hernandez-Vicente A, Pascual-Figal DA; clinical trial REMOVE researches. Withdrawal of drug therapy in responders to cardiac resynchronization therapy: rationale and design of the REMOVE trial. Rev Esp Cardiol (Engl Ed). 2024 Oct;77(10):851-858. doi: 10.1016/j.rec.2024.02.021. Epub 2024 May 1. English, Spanish. PMID 38701881